CLINICAL TRIAL: NCT05864664
Title: Comparing Removal of Ankle Implants/ Hardware Using the Wide-awake Local Anesthesia no Tourniquet (WALANT) Technique Versus General Anesthesia.
Brief Title: Safety and Efficacy of Wide Awake Local Anesthesia no Tourniquet Technique (WALANT) in Ankle Removal of Implant Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ali Lari (Other Government)
Responsible Party: Sponsor-Investigator, Ali Lari, Dr Ali Lari - MB BCh BAO, Kuwait Institute for Medical Specialization
Organization: Kuwait Institute for Medical Specialization (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2027
Record Dates: First submitted 2022-08-16; First posted 2023-05-18 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Safety Issues; Post Operative Pain; Local Anesthetic Complication
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, therapeutic, comparative, randomized controlled ?
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WALANT procedure (Experimental): Patient awake with no form of sedation or analgesia
  A mixture of lidocaine, adrenaline, normal saline, bicarbonate is used to get 40-50ml solution Injection is performed around incision site - superficial to deep including periosteum Incision is performed in the normal fashion Plate and screws are removed and incision is closed
  Interventions: Procedure: Wide awake local anaesthesia no tourniquet technique
- General anesthesia (Active Comparator): The surgery is performed in the standard fashion. The patient received general anesthesia The surgery is performed normally and the plate/screws are removed
  Interventions: Procedure: Wide awake local anaesthesia no tourniquet technique

INTERVENTIONS:
Procedure: Wide awake local anaesthesia no tourniquet technique — Patient awake with no form of sedation or analgesia
  * A mixture of lidocaine, adrenaline, normal saline, bicarbonate is used to get 40-50ml solution
  * Injection is performed around incision site - superficial to deep including periosteum
  * Incision is performed in the normal fashion
  * Plate and screws are removed and incision is closed

SUMMARY:
Safety and efficacy of wide awake local anesthesia no torniquet technique (WALANT) in ankle surgery. Studying risks and benefits from WALANT compared to general anesthesia . WALANT expected to decrease in intraoperative/post operative pain at the surgical site and decrease hospital time .

ELIGIBILITY:
Inclusion Criteria:

* Age: >18
* Previous ORIF for:
* Unimalleolar fractures
* Bimalleolar fractures
* Trimalleolar fractures

Exclusion Criteria:

* Allergy to local anesthesia
* Psychiatric diagnosis including: affect disorders, uncooperative
* Severe cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the patient's maximum pain intraoperatively at the surgical site | Intraoperative
  Visual analogue pain scale - VAS
Blood loss | Intraoperative
  Amount cc

CONTACTS AND LOCATIONS:
Overall Officials: Ali Jarragh, MD FRCS.C, Principal Investigator — Kuwait University
Locations (1):
- AlRazi Orthopedic Hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided